CLINICAL TRIAL: NCT03014713
Title: Effect of Dexmedetomidine Combined With Dezocine and Flubiprofen for Postoperative Intravenous Patient Controlled Analgesia After Colorectal Surgery
Brief Title: Effect of Dexmedetomidine for Postoperative Intravenous Patient Controlled Analgesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weifeng Tu (Other)
Responsible Party: Sponsor-Investigator, Weifeng Tu, Chief Physician, Guangzhou General Hospital of Guangzhou Military Command
Organization: Guangzhou General Hospital of Guangzhou Military Command (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Dexmedetomidine PCA
Record Dates: First submitted 2017-01-03; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Patient-Controlled Analgesia
Keywords: Dexmedetomidine; Dezocine; Flubiprofen; Analgesia; Colorectal Surgery
MeSH Terms: conditions — Agnosia | interventions — dezocine; Flurbiprofen; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): Patients in this group receive intravenous Patient-Controlled Analgesia(PCA) pump after surgery.The intravenous PCA protocol is dezocine 0.01mg/kg/h,flubiprofen 0.05mg/kg/h.
  Interventions: Drug: Dezocine; Drug: Flubiprofen
- Dexmedetomidine Group (Experimental): Patients in this group receive intravenous Patient-Controlled Analgesia(PCA) pump after surgery.The intravenous PCA protocol is dezocine 0.01mg/kg/h,flubiprofen 0.05mg/kg/h,dexmedetomidine 0.1μg/kg/h.
  Interventions: Drug: Dezocine; Drug: Flubiprofen; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dezocine — Dezocine 0.01mg/kg/h intravenous administration during the first two days after surgery.
Drug: Flubiprofen — Flubiprofen 0.5mg/kg/h intravenous administration during the first two days after surgery.
Drug: Dexmedetomidine — Dexmedetomidine 0.1μg/kg/h intravenous administration during the first two days after surgery.
  Arms: Dexmedetomidine Group

SUMMARY:
The purpose of this study is to explore the effectiveness of dexmedetomidine as an adjunctive analgesic, combined with dezocine and flubiprofen, used in intravenous Patient-Controlled Analgesia (PCA) after open colorectal surgery.

DETAILED DESCRIPTION:
Dexmedetomidine is a selective alpha-2 adrenoceptor agonist, which has been demonstrated to have anaesthetic, sedative and analgesic-sparing effects. Besides, Dexmedetomidine has been reported to cause sedative effects and reduce opioid requirements in the perioperative period. Many studies had been conducted to reduce the side effect of opioid analgesic. The current trend of reducing opioid analgesic side effect is direct combination of other drugs in PCA. The advantages of this method are convenient in clinical use and preventive for side effects.

In this study, 50 patients who is undergoing elective colorectal surgery will be randomly allocated into two groups (Control group and Dexmedetomidine group). Patients in both groups will be given a patient-controlled analgesia (PCA) pump in post anesthetic recovery unit (PACU) after surgery.

The PCA protocol of Control group is dezocine 0.6mg/kg, flubiprofen 3mg/kg, diluted into 120ml and administer at a background infusion of 2ml/h, and a bolus of 2ml, with a lock-out of 15min. The PCA protocol of Dexmedetomidine group is dezocine 0.6mg/kg, flubiprofen 3mg/k and dexmedetomidine 6μg/kg diluted into 120ml and administer at a background infusion of 2ml/h, and a bolus of 2ml, with a lock-out of 15min.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists(ASA) Ⅰ-Ⅱ patient undergoing open colorectal surgery
2. Written informed consent from the patient or the relatives of the participating patient.
3. BMI:18～30kg/m2

Exclusion Criteria:

1. Mental illness or cannot communicate.;
2. A second operation during the study;
3. Slow-type arrhythmias or hypotension;
4. Lung infection or sleep apnea syndrome;
5. Renal failure;
6. Alcohol or drug abuse;
7. Already taking gabapentin, pregabalin, benzodiazepin or antidepression drug;
8. Long-term use of analgesics,sedatives or non steroidal anti-inflammatory drugs history;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Dezocine consumption by patient-controlled analgesia | At 24 hours after surgery
  The total consumption of dezocine during 24 hours after surgery are recorded.
Change in pain score | At 0, 2, 4, 8, 24, 48 and 72 hours after surgery
  Pain scores at rest and movement are evaluated with a numeric rating scale (NRS).

SECONDARY OUTCOMES:
Change in ramsay sedation score | At 0, 2, 4, 8, 24, 48 and 72 hours after surgery
  Measure sedation level by using ramsay sedation score
The incidence rates of postoperative nausea and vomiting (PONV) | At 24 hours after surgery
  Measure whether nausea and vomiting exist and the level of severity.

CONTACTS AND LOCATIONS:
Overall Officials: Weifeng Tu, PhD, Principal Investigator — Guangzhou General Hospital of Guangzhou Military Command
Locations (1):
- Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Bellon M, Le Bot A, Michelet D, Hilly J, Maesani M, Brasher C, Dahmani S. Efficacy of Intraoperative Dexmedetomidine Compared with Placebo for Postoperative Pain Management: A Meta-Analysis of Published Studies. Pain Ther. 2016 Jun;5(1):63-80. doi: 10.1007/s40122-016-0045-2. Epub 2016 Feb 10. PMID 26861737
- [Background] Ge DJ, Qi B, Tang G, Li JY. Intraoperative Dexmedetomidine Promotes Postoperative Analgesia and Recovery in Patients after Abdominal Hysterectomy: a Double-Blind, Randomized Clinical Trial. Sci Rep. 2016 Feb 23;6:21514. doi: 10.1038/srep21514. PMID 26903197
- [Background] Jessen Lundorf L, Korvenius Nedergaard H, Moller AM. Perioperative dexmedetomidine for acute pain after abdominal surgery in adults. Cochrane Database Syst Rev. 2016 Feb 18;2(2):CD010358. doi: 10.1002/14651858.CD010358.pub2. PMID 26889627